CLINICAL TRIAL: NCT04923646
Title: Primers to Improve Adherence to Annual CRC Screening Among Veterans: A Randomized Control Trial
Brief Title: Veteran Primers for CRC Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alaina Mori, Staff Physician, VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: FIT1
Record Dates: First submitted 2021-05-19; First posted 2021-06-11 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
Keywords: Cancer screening; Behavioral economics; Adherence
MeSH Terms: conditions — Colorectal Neoplasms | interventions — DNA Primers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Primer
  Interventions: Other: Primer
- Control (No Intervention): No Primer

INTERVENTIONS:
Other: Primer — Mailed postcard notifying Veteran of upcoming FIT kit for annual CRC screening.
  Arms: Active

SUMMARY:
This is a prospective, randomized controlled trial that will evaluate the effectiveness of primer postcards sent two weeks prior to the mailing of a FIT kit in improving adherence to annual CRC screening. This project is for the purpose of quality improvement and has been designated as non-research by the VHA Office of Primary Care, Improvement & Innovation (VHA Program Guide 1200.21).

DETAILED DESCRIPTION:
Veterans eligible for enrollment into the trial will be randomized in a 1:1 allocation using permuted block randomization (with random block sizes of 4 and 8) to the following interventions:

1. Active arm: Primer

   1. Intervention Type: Other
   2. Intervention Description: Mailed postcard notifying Veteran of upcoming FIT kit receipt for annual CRC screening
2. Control arm: No primer a. Intervention Type: No intervention

Randomization will be stratified within arms by prior screening status (prior screener vs. never screener)

Our primary outcome of interest is the return rate at three months post randomization. Our secondary outcome of interest is the return rate at six months post randomization. Enrollment in the trial will occur between May 1, 2021 and January 1, 2022.

ELIGIBILITY:
Eligible participants are automatically enrolled in this project. We are unable to enroll participants upon request.

Inclusion criteria:

* Veteran
* Assigned to a primary care provider at the VA Puget Sound as of January 1, 2021
* At least 1 year of prior data available (evidence of at least one outpatient visit)
* Due for annual colorectal (CRC) screening

Exclusion criteria:

* Not scheduled for either a screening or diagnostic colonoscopy within the 12 weeks from assessment.
* Not currently receiving hospice care
* No record of recent death in the administrative data.
* No history of CRC or history of prior colectomy.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2404 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Return proportion | 3 months
  Percent of returned FIT tests

SECONDARY OUTCOMES:
Return proportion | 6 months
  Percent of returned FIT tests

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Reddy, MD, Principal Investigator — VA Puget Sound Health Care System; Stefanie Deeds, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No